CLINICAL TRIAL: NCT03764280
Title: An Open-Label, Randomized, Two-Way, Parallel Study to Compare the Efficacy of MDI Treatment With Physician Adjusted and Optimization Algorithm Adjusted Basal-Bolus Parameters in Children and Adolescents With Type 1 Diabetes at a Diabetes Camp
Brief Title: The Efficacy of MDI Treatment With an Optimization Algorithm Adjusting Basal-Bolus Parameters in Children and Adolescents With Type 1 Diabetes at a Diabetes Camp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDI Optimization Algorithm
Record Dates: First submitted 2018-06-27; First posted 2018-12-05 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Diabete Mellitus; Diabetes Mellitus, Type 1
Keywords: Multiple Daily Injections; type 1 diabetes; pediatrics; optimization algorithm
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin, Short-Acting

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, two-way, parallel study to compare the glucose control between physician adjusted basal-bolus parameters and our computer basal-bolus optimizing algorithm. Children and adolescent type 1 diabetes patients at Camp Carowanis, a camp for diabetes, will be enrolled in the study, where they will randomly undergo one of two interventions:
  1. MDI with Physician Adjusted Basal-Bolus Parameters
  2. MDI with Basal-Bolus Optimization Algorithm Adjusted Basal-Bolus Parameters (OA)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MDI with Physician Adjusted Basal-Bolus Parameters (No Intervention): Participants will be wearing the Freestyle Libre glucose sensor (Abbott Diabetes Care). Participants will undergo their conventional multiple daily injection (MDI) therapy.
- MDI with Basal-Bolus Optimization Algorithm (Experimental): Participants will be wearing the Freestyle Libre glucose sensor (Abbott Diabetes Care). Once daily, the data from the glucose sensor and injection information will be entered into a computer and the optimization algorithm will be run. Once daily, participants' parameters may be changed based on the algorithm's recommendations.
  Interventions: Other: Multiple Daily Injections: Slow acting insulin and Rapid acting insulin

INTERVENTIONS:
Other: Multiple Daily Injections: Slow acting insulin and Rapid acting insulin — Multiple daily injections (MDI) therapy involves four or more daily insulin injections. Once or twice daily, a long acting insulin is injected as a basal dose. These long acting insulins are designed to dissipate slowly and evenly into the bloodstream for 24 to 36 hours following injection. This basal injection aims to mimic the physiological healthy basal insulin released from a healthy pancreas all day. Furthermore, multiple insulin bolus doses are injected at every meal each day using rapid or short acting insulin. These injections are administered before meals and are calculated using patients' ICRs and meal carbohydrate quantities.
  Arms: MDI with Basal-Bolus Optimization Algorithm

SUMMARY:
Our lab at McGill University has developed an optimization algorithm for T1D MDI patients that estimates optimal basal-bolus parameters (basal injections and insulin-to-carbohydrate ratios) using glucose sensor data and insulin dosing data over several days. The algorithm examines daily glucose, insulin, and meal data to make changes in patients' basal injections and ICRs. The investigators hope that this algorithm will be able to optimize the patients' individual basal injections and ICRs in order to improve glycemic control.

DETAILED DESCRIPTION:
The objective of this project is to compare our basal-bolus optimization algorithm with physician adjusted basal-bolus parameters using a randomized parallel clinical trial in children and adolescents at a Camp Carowanis. The investigators hypothesize that using this optimization algorithm will be non-inferior to the physician-adjusted basal-bolus parameters regarding time spent in target glucose range (3.9 mmol/L - 10mmol/L).

Between 40 and 68 children and adolescent type 1 diabetes patients undergoing MDI treatment at Camp Carowanis will randomly undergo one of two interventions:

1. MDI with Physician Adjusted Basal-Bolus Parameters: Participants will be wearing the Freestyle Libre glucose sensor (Abbott Diabetes Care). Participants will undergo their conventional multiple daily injection (MDI) therapy. At breakfast, the research team will download the sensor data. Camp physicians will review each participant's sensor and insulin data and make changes to their parameters based on their clinical judgement, as they would for all campers, regardless of study participation. These new parameters will be entered into the patient's camp file.
2. MDI with Basal-Bolus Optimization Algorithm Adjusted Basal-Bolus Parameters: Participants will be wearing the Freestyle Libre glucose sensor (Abbott Diabetes Care). At breakfast, the data from the glucose sensor and injection information will be entered into a computer and the optimization algorithm will be run. Camp physicians will review the algorithm's recommendations before they are entered into the patient's camp file.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 8 and 18 years old.
2. Clinical diagnosis of type 1 diabetes for at least 12 months. The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
3. Undergoing multiple daily injection therapy.
4. HbA1c ≤ 11%.

Exclusion Criteria:

1. Serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
2. Failure to comply with the study protocol or with team's recommendations.
3. Injection of isophane insulin (NPH) or any intermediate-acting insulin
4. More than one injection of slow-acting insulin per day.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Percentage of time of sensor glucose levels spent in target range (defined to be between 3.9 mmol/L and 10.0 mmol/L). | the last 7 days of the study.

SECONDARY OUTCOMES:
Percentage of time of sensor glucose levels spent: | last 7 days of the study
  a. between 3.9 and 7.8 mmol/L; b. between 3.9 and 10 mmol/L; c. below 3.9 mmol/L; d. below 3.3 mmol/L; e. below 2.8 mmol/L; f. above 7.8 mmol/L; g. above 10 mmol/L; h. above 13.9 mmol/L; i. above 16.7 mmol/L.
Percentage of overnight time (23:00-7:00) of sensor glucose levels | last 7 days of the study
  a. between 3.9 and 7.8 mmol/L; b. between 3.9 and 10 mmol/L; c. below 3.9 mmol/L; d. below 3.3 mmol/L; e. below 2.8 mmol/L; f. above 7.8 mmol/L; g. above 10 mmol/L; h. above 13.9 mmol/L; i. above 16.7 mmol/L.
Percentage of daytime (7:00-23:00) of sensor glucose levels | last 7 days of the study
  a. between 3.9 and 7.8 mmol/L; b. between 3.9 and 10 mmol/L; c. below 3.9 mmol/L; d. below 3.3 mmol/L; e. below 2.8 mmol/L; f. above 7.8 mmol/L; g. above 10 mmol/L; h. above 13.9 mmol/L; i. above 16.7 mmol/L.
Standard deviation of glucose levels as a measure of glucose variability | last 7 days of the study
Total insulin delivery. | last 7 days
Mean sensor glucose level during | last 7 days
  a. the overall study period; b. the daytime period; c. overnight period.
Number of participants experiencing hypoglycemia requiring oral treatment during | last 7 days
  a. the overall study period; b. the daytime period; c. overnight period.

CONTACTS AND LOCATIONS:
Locations (1):
- Camp Carowanis, Sainte-Agathe-des-Monts, Quebec, Canada